CLINICAL TRIAL: NCT06814275
Title: Project ARTEMIS: A Mechanistic Clinical Trial of Neuroimmune Pathways.
Brief Title: Project neuroARTEMIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Florida International University (Other); National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00117907; 1R01DA061952-01 (NIH)
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Stimulant Use; Human Immunodeficiency Virus (HIV); Depression
Keywords: HIV; Stimulant use; substance abuse; chronic stress
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Depression; Substance-Related Disorders | interventions — Anti-Retroviral Agents

STUDY DESIGN:
Intervention Model Description: This study will utilize two treatment arms in which participants are randomized using a 2:1 allocation. Arm A will receive the ARTEMIS intervention immediately following their baseline visit. Arm B will be considered a wait-list control, being offered the ARTEMIS intervention after a 6-month delay.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARTEMIS (Active Comparator): Participants in this arm will receive the ARTEMIS intervention immediately following randomization.
  Interventions: Behavioral: ARTEMIS; Behavioral: Contingency management for Antiretroviral (ARV) adherence
- Waitlist Control (WLC) (Other): Participants in the WLC arm will be offered the ARTEMIS intervention after the final (6-month) follow-up.
  Interventions: Behavioral: Contingency management for Antiretroviral (ARV) adherence

INTERVENTIONS:
Behavioral: ARTEMIS — The ARTEMIS intervention includes 5 sessions delivered individually over Zoom across 3 months. The intervention teaches 9 positive affect skills: noting and capitalizing on positive events, gratitude journaling, formal and informal mindfulness, positive reappraisal and problem solving coping skills training, focusing on personal strengths, setting achievable goals, and small acts of kindness. Each session consists of a didactic portion with in vivo skills practice, and participants are asked to complete daily home practice of the skills between sessions.
  Arms: ARTEMIS
Behavioral: Contingency management for Antiretroviral (ARV) adherence — All participants will received the contingency management (CM) intervention to support ARV adherence. They will use the Spotlight by Scene Health platform, a HIPAA-compliant mHealth application for directly observed therapy, to upload videos of ART adherence. The app records and uploads time-stamped videos of medication doses, which staff verify asynchronously. Participants will be paid for each verified dose and receive a weekly bonus if they complete 6 doses.

SUMMARY:
The purpose of this research is to understand how chronic stress affects the way our brain and immune systems function, and in turn how this affects the way people feel, think, and behave. By learning more about how these processes work, the hope is to be able to develop better treatments to help with problems like depression and substance use. This study is intended for individuals that are HIV positive, currently taking prescription antiretroviral medications, and use stimulants. Through this intervention, the aim is to determine if this positive affect intervention can lead to reductions in stimulant use and depressed mood.

DETAILED DESCRIPTION:
Participants who meet initial eligibility criteria will complete a baseline assessment that includes psychosocial and behavioral measures, biospecimen collection, and an MRI brain scan. Participants will then be randomized to either: 1) ARTEMIS; or 2) a waitlist control (WLC) condition. ARTEMIS participants will receive 5 sessions delivered individually over Zoom across 3 months. All participants (including WLC) will receive contingency management (CM) for antiretroviral therapy (ART) adherence to support sustained viral suppression over the active phase of the trial. During the intent-to-treat period, assessments at 3- and 6-month follow-ups will characterize changes in neural activity (assessed via fMRI) and conserved transcriptional response to adversity (CTRA) leukocyte signaling (assessed via RNA sequencing) as plausible mediators of behavioral outcomes following ARTEMIS. WLC participants will be offered the ARTEMIS intervention after a 6-month delay.

ELIGIBILITY:
Inclusion Criteria:

* 18-59 years old
* Weekly use of stimulants reported in the past month or a score of 4 or more on the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST)
* Confirmed HIV diagnosis
* Current receipt of daily oral antiretroviral therapy (ART) medication
* English fluency/literacy

Exclusion Criteria:

* Acute brain infection (e.g., neurosyphilis, toxoplasmosis)
* Acutely symptomatic bipolar I or psychotic disorder
* Prescription for immunomodulatory medications or other immunotherapy
* Any MRI contraindications
* If applicable, on antidepressant medication regimen for at least 2 months

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 189 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Neural Functional Connectivity | Month 3
  Functional connectivity (FC) will be derived from the the resting-state functional MRI data. Using a theory-driven, seed-based approach, the 4D time series [average blood oxygenation level dependent (BOLD) signal across voxels] will be extracted from a priori seeds in the reward network (i.e., nucleus accumbens, subgenual anterior cingulate cortex, medial orbitofrontal cortex). Normalized Z-scores will be calculated for FC between regions of interest. These analyses will control for baseline FC.
Neural Activation | Month 3
  The Monetary Incentive Delay Task will be used to probe neural activation to reward processing, using an event-level design. Blood oxygenation level dependent (BOLD) activation will be modeled as a canonical hemodynamic response function specified at stimulus onset. Event epochs that are time locked to the onset of each trial will be extracted from the overall time series. Random-effects general linear model will be used to calculate statistical parametric maps reflecting the probability that a voxel is activated as a function of the experimental task. The primary analysis will focus on nucleus accumbens and ventromedial prefrontal cortex activity as regions of interest (ROI). Mean beta values will be averaged across all voxels in each ROI. These analyses will control for baseline activation levels.

SECONDARY OUTCOMES:
Change in Frequency of Stimulant Use | 3 and 6 month follow-ups
  Utilizing a Timeline Follow-back, days of stimulant use in past 30 will be assessed. Stimulants will include methamphetamine, other amphetamines, cocaine, and other stimulants. Change in use from baseline will be examined.
Depression Scores | 3 and 6 month follow-ups
  Depression symptom severity, measured via (CES) Center for Epidemiologic Studies Depression Scale. This assessment is a 20 item assessment with each item being assigned a value of 0-3. Higher scores are indicative of depression. The total score is calculated by calculating the sum of 20 items. Scores range from 0-60, with higher scores meaning greater depressive symptoms. We will examine change from baseline.
CTRA Leukocyte Signaling | Baseline, Month 3, Month 6
  RNA sequencing (RNAseq) of peripheral blood mononuclear cells (PBMCs) will be conducted for analysis of differential gene expression, detection of low expressed genes, allele specific expression analysis, and splice variants. Gene expression values will be log2-transformed and pre-specified sets of inflammatory and Type I interferon genes will be combined into a single-number CTRA indicator (53-gene contrast score).
Change in Peripheral Inflammation | 3 and 6 month follow-ups
  Plasma samples will undergo multiplexed analysis for key inflammatory mediators: CRP, TNF-a, IFN-g, IL-1b, IL-6, CXCL10, and CCL2. Single-enzyme-linked immunoabsorbent assays (ELISAs) will be performed for sCD14 and sCD163. We will examine changes in concentration from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Christina S Meade, PhD, Principal Investigator — Wake Forest University Health Sciences; Adam W Carrico, PhD, Principal Investigator — Florida International University
Locations (1):
- Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual-level phenotypic, clinical, genomic, and neuroimaging data for all research subjects will be preserved and deposited in designated NIH-supported repositories for sharing broadly with the scientific community (described below). While identifiers will be collected, all data will be de-identified prior to deposit into any repository. Shared data will include raw and processed files for genomic and neuroimaging data. Recruitment progress and final results will be documented at ClinicalTrials.gov. The sources of data include clinical interviewing, computerized questionnaires, neuropsychological testing, biological sampling (blood and urine), MRI neuroimaging, and medical record review. The final dataset from this project will also include data on demographic factors (including biological variables) and clinical variables such as HIV disease characteristics.
Supporting Information: Study Protocol, ICF
Time Frame: The investigators will lock the data until the primary analyses are completed and accepted for publication, after which the investigators will make the data as widely available as possible. Data and supporting documentation will be prepared for deposit in the appropriate repositories in Years 4-5 of the project, with deposit occurring in the final quarter of Year 5 (Q4 2029).
Access Criteria: All data for all research subjects will be preserved and deposited in designated NIH-supported repositories for sharing broadly with the scientific community. Anyone with access to these repositories will have access to the deidentified data from this project.